CLINICAL TRIAL: NCT00775268
Title: A Pilot Study of 18F Fluorothymidine (FLT) PET/CT in Lymphoma
Brief Title: 18F- Fluorothymidine to Evaluate Treatment Response in Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Esther Mena, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 080200; 08-C-0200
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Lymphoma
Keywords: 18F-Fluorothymidine; PET/CT; FLT; Lymphoma; FDG
MeSH Terms: conditions — Lymphoma | interventions — Biopsy; Tomography, X-Ray Computed; Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group A - Participants Scanned at Baseline & After Chemotherapy (Experimental): Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) PET/CT scans at baseline, after 2 courses of chemotherapy, and after completion of chemotherapy. Patients with residual FDG-positive mass after completion of therapy may be enrolled in group B.
  Interventions: Diagnostic Test: fluorodeoxyglucose F 18 Positron Emission Tomography and computed tomography; Other: [3'-deoxy-3'-[F-18] fluorothymidine; Procedure: computed tomography
- Group B - Participants Scanned in the Evaluation of Residual Masses After Therapy (Experimental): Patients who have completed treatment in whom FDG-PET shows a remaining tumor mass undergo an FLT PET/CT scan . Patients also undergo a biopsy or fine-needle aspiration, if clinically indicated.
  Interventions: Procedure: Biopsy; Diagnostic Test: fluorodeoxyglucose F 18 Positron Emission Tomography and computed tomography; Other: [3'-deoxy-3'-[F-18] fluorothymidine; Procedure: computed tomography; Procedure: fine-needle aspiration

INTERVENTIONS:
Procedure: Biopsy — Biopsy taken
  Arms: Group B - Participants Scanned in the Evaluation of Residual Masses After Therapy
Diagnostic Test: fluorodeoxyglucose F 18 Positron Emission Tomography and computed tomography — Imaging
Other: [3'-deoxy-3'-[F-18] fluorothymidine — Undergo scans
Procedure: computed tomography — Undergo scans
Procedure: fine-needle aspiration — sample collected
  Arms: Group B - Participants Scanned in the Evaluation of Residual Masses After Therapy

SUMMARY:
Background:

* Positron emission tomography (PET) uses radioactive substances called radiotracers to locate areas of cancer in the body. For this test, the patient is given an injection of the radiotracer and lies in a large donut-shaped scanner that detects where in the body the radioactivity accumulates. Computed tomography (CT) scans use low dose x-rays that help to better localize where the radioactive tracer is concentrating. PET/CT scans are usually done in lymphoma patients before treatment starts and at the end of treatment to evaluate the response to therapy.
* PET scans typically use a sugar-like radioactive tracer called fluorodeoxyglucose (FDG) and low-dose x-rays. Sometimes, however, FDG PET scans show what looks like active disease and presence of a mass after chemotherapy even when there are no live cancer cells. Doctors have particular problems in evaluating response to treatment when this happens because they can't tell if the mass is active cancer or just dead tumor cells.
* An experimental radiotracer called 18F- Fluorothymidine (FLT) has high uptake in active tumor cells and may be better able to evaluate treatment response.

Objectives:

- To test the use of FLT PET/CT imaging in assessing treatment response in patients with lymphoma.

Eligibility:

- Patients 18 years of age or older who are enrolled in a lymphoma therapy study at the National Institutes of Health (NIH) Clinical Center or in the Cancer and Leukemia Group B (CALGB) 50330 study at another location.

Design:

- There are two arms in this study:

* The first arm evaluates FLT as an early predictor of tumor response to therapy. Patients are imaged with FLT and FDG PET before starting treatment, following two cycles of therapy and after treatment ends.
* The second arm evaluates the ability of FLT to distinguish if a mass that remains after treatment has viable cancer or dead tissue. Patients who have completed treatment and in whom FDG PET shows a remaining tumor mass are imaged with FLT PET. Following the scan, the tumor is biopsied for verification.

DETAILED DESCRIPTION:
Background:

* 3-deoxy-3-18F-fluorothymidine (FLT) positron emission tomography (FLT PET)/Compute tomography (CT) has been shown to correlate with the rate of cellular/tumor proliferation.
* The Imaging Subcommittee of the International Harmonization Project in Lymphoma recommends performing fluorodeoxyglucose (FDG) positron emission tomography (PET) at least 3 weeks, and preferably 6-8 weeks after chemotherapy or chemoimmunotherapy and 8-12 weeks after radiation or chemoradiation therapy due to high FDG accumulation in inflammatory tissues.
* FLT uptake in inflammatory lesions is less prominent than FDG and it is likely that FLT PET/CT can better differentiate inflammation from tumor.
* FLT PET/CT imaging is expected to better differentiate between treatment induced inflammation and malignancy and should enable early prediction of therapeutic response.
* FLT PET/CT imaging is expected to differentiate between residual inflammatory residual masses from residual malignancy and therefore guide appropriate treatment.

Primary Objectives:

* To estimate the diagnostic accuracy of FLT PET/CT as an early indicator of complete response to therapy in B and T cell lymphoma.
* To estimate the diagnostic accuracy of FLT PET/CT in the evaluation of residual masses after therapy.

Eligibility:

* Participant must be enrolled in a lymphoma therapy study at the National Institutes of Health (NIH) Clinical Center OR be enrolled in the CALGB 50303 study at another site OR undergoing a new course of treatment of lymphoma at another facility. The National Cancer Institute (NCI) Laboratory of Pathology will confirm diagnosis for subjects enrolled at all CALGB study sites.
* Participants must have a clinical course consistent with lymphoma and have available documentation of lymphoma from either the NCI or from an outside pathology laboratory.
* Subjects enrolling in the early response arm must undergo baseline FLT PET prior to receiving a new course of lymphoma therapy.
* Subjects enrolling in the residual mass evaluation arm can be enrolled at the time the FDG avid residual mass is discovered (i.e. no pre-therapy FLT image is required).
* Subjects can enroll in both arms of the study.
* Participant must be 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 or 1.
* Serum glutamic-oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase (SGPT) less than 5 times upper limit of normal (ULN).
* bilirubin less than or equal to 2 times ULN.

Design:

There are 2 arms in this study

* The first arm will assess FLT as an early predictor of tumor response to therapy (treatment naive or recurrent disease). Subjects are imaged with FLT and FDG PET pre-therapy, following 2 cycles of therapy and post therapy.
* The second arm will assess lymphoma patients with FDG PET positive residual mass. Subjects are imaged with FLT PET prior to standard of care biopsy of residual mass. If initial FDG PET data is not available in Digital Imaging and Communications in Medicine (DICOM) format or is of suboptimal image quality, a repeat FDG PET/CT at the study site may be required.

  * We will accrue 70 participants (40 in the early response arm and 30 in the residual mass arm) to this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participant must be enrolled in a lymphoma therapy study at the National Institutes of Health (NIH) Clinical Center OR be enrolled in the Cancer and Leukemia Group B (CALGB) 50303 study at another site OR undergoing a new course of treatment of lymphoma at another facility.

Participants must have a clinical course consistent with lymphoma and have available documentation of lymphoma from either the National Cancer Institute (NCI) or from an outside pathology laboratory.

Participant must be 18 years or older.

Eastern Cooperative Oncology Group (ECOG) Performance score of 0 or 1.

Ability to provide informed consent. All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

For subjects enrolling in early response arm

* Must be enrolled in CALGB 50303 or a lymphoma therapy study at the NIH Clinical Center or undergoing a new course of treatment of lymphoma at another facility
* Must not have begun lymphoma therapy for this tumor occurrence/ relapse
* Prior completed therapy does NOT affect eligibility

For subjects enrolling in the residual FDG avid mass arm

* Must have a residual (18)F-fluorodeoxyglucose (FDG) positron emission tomography (PET) positive mass greater than equal to 1cm, with uptake greater than that of mediastinal blood pool.
* Participant will undergo a repeat FDG PET/CT scan if the original FDG/PET imaging performed at an outside institution is not of adequate imaging quality for subjects enrolling in the residual FDG mass arm.

EXCLUSION CRITERIA:

Known allergy to fluorothymidine.

Participants for whom enrollment would significantly delay (greater than 2 weeks) the scheduled standard of care therapy.

Participants with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results are excluded.

Participants with severe claustrophobia not relieved by oral anxiolytic medication or patients weighing greater than 136 kg (weight limit for scanner table).

Other medical conditions deemed by the Principal Investigator (PI) or associates to make the patient ineligible for protocol procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09-29 (Actual); Primary Completion 2014-10-23 (Actual); Study Completion 2014-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Mena, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Walter Reed National Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spaepen K, Stroobants S, Dupont P, Vandenberghe P, Thomas J, de Groot T, Balzarini J, De Wolf-Peeters C, Mortelmans L, Verhoef G. Early restaging positron emission tomography with ( 18)F-fluorodeoxyglucose predicts outcome in patients with aggressive non-Hodgkin's lymphoma. Ann Oncol. 2002 Sep;13(9):1356-63. doi: 10.1093/annonc/mdf256. PMID 12196360
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Scanned at Baseline & After Chemotherapy: Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scans at baseline, after 2 courses of chemotherapy, and after completion of chemotherapy. Patients with residual FDG-positive mass after completion of therapy may be enrolled in group B.
  Fluorodeoxyglucose F 18: Undergo scans [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans
- Participants Scanned in the Evaluation of Residual Masses After Therapy: Patients undergo a 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scan in the evaluation of FDG-positive residual masses after therapy. Patients also undergo a biopsy or fine-needle aspiration, if clinically indicated.
  Biopsy: Biopsy taken [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans fine-needle aspiration: sample collected
Period: Baseline
Arm/Group | Participants Scanned at Baseline & After Chemotherapy | Participants Scanned in the Evaluation of Residual Masses After Therapy
Started | 9 | 22
Completed | 8 | 21
Not Completed | 1 | 1
Not completed — Drug not synthesize dose | 1 | 0
Not completed — Not treated-ineligible per CT | 0 | 1
Period: After 2 Cycles
Arm/Group | Participants Scanned at Baseline & After Chemotherapy | Participants Scanned in the Evaluation of Residual Masses After Therapy
Started | 8 | 0 (These 21 patients were not scanned after 2-cycles in this Arm. They were only scanned at baseline.)
Completed | 7 | 0
Not Completed | 1 | 0
Not completed — Participant refused to be scanned further | 1 | 0
Period: After Completion
Arm/Group | Participants Scanned at Baseline & After Chemotherapy | Participants Scanned in the Evaluation of Residual Masses After Therapy
Started | 7 | 0
Completed | 6 | 0
Not Completed | 1 | 0
Not completed — Participant missed scan appointment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Scanned at Baseline & After Chemotherapy | Participants Scanned in the Evaluation of Residual Masses After Therapy | Total
Number analyzed (Participants) | 9 | 22 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 18 | 26
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (13.0) | 48.0 (17.3) | 48.4 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15
  Male | 6 | 10 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 21 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 9 | 17 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 22 | 31
Diagnosis [Number; unit: participants]
  Non-Hodgkin's Lymphoma | 6 | 17 | 23
  Hodgkin's Lymphoma | 3 | 5 | 8
Residual Mass Size [Number; unit: cm] — Population: Measurement of lesions was not required to qualify for scanning in the first Arm/Group. These are 9 different patients scanned before starting chemo (these patients have not Residual Masses). And Note: 21 patients were not scanned after 2-cycles in the Participants Scanned in the Evaluation of Residual Masses After Therapy Arm. They were only scanned at baseline.
  cm
    Patient 1-Right hilum lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 1-Right hilum lymph node |  | 2.4 | 2.4
    Patient 2-Superior mediastinal lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 2-Superior mediastinal lymph node |  | 2.4 | 2.4
    Patient 3-Lumbar vertebrae: number analyzed (Participants) | 0 | 1 | 1
    Patient 3-Lumbar vertebrae |  | 2.5 | 2.5
    Patient 4-Right pelvic mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 4-Right pelvic mass |  | 9.0 | 9.0
    Patient 5-Intercostal soft tissue mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 5-Intercostal soft tissue mass |  | 2.3 | 2.3
    Patient 6-Right cervical lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 6-Right cervical lymph node |  | 3.7 | 3.7
    Patient 7-Anterior mediastinal mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 7-Anterior mediastinal mass |  | 2.7 | 2.7
    Patient 8-Anterior mediastinal mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 8-Anterior mediastinal mass |  | 6.8 | 6.8
    Patient 9-Internal right iliac lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 9-Internal right iliac lymph node |  | 2.2 | 2.2
    Patient 10-Right pelvic mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 10-Right pelvic mass |  | 2.2 | 2.2
    Patient 11-Right paratracheal lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 11-Right paratracheal lymph node |  | 2.0 | 2.2
    Patient 12-Left inguinal lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 12-Left inguinal lymph node |  | 1.6 | 1.6
    Patient 13-Left axilla lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 13-Left axilla lymph node |  | 3.0 | 3.0
    Patient 14-Gastrohepatic lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 14-Gastrohepatic lymph node |  | 2.8 | 2.8
    Patient 15-Right posterior thigh mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 15-Right posterior thigh mass |  | 2.5 | 2.5
    Patient 16-Left abdominal mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 16-Left abdominal mass |  | 8.0 | 8
    Patient 17-Left suprarenal mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 17-Left suprarenal mass |  | 4.3 | 4.3
    Patient 18-Splenic mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 18-Splenic mass |  | 2.3 | 2.3
    Patient 19-Right paraaortic lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 19-Right paraaortic lymph node |  | 2.7 | 2.7
    Patient 20-Right hilum lymph node: number analyzed (Participants) | 0 | 1 | 1
    Patient 20-Right hilum lymph node |  | 1.6 | 1.6
    Patient 21-Mesenteric mass: number analyzed (Participants) | 0 | 1 | 1
    Patient 21-Mesenteric mass |  | 5.2 | 5.2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Presence/Absence of Abnormal 18F- Fluorothymidine (FLT) Uptake, and Positive/Negative Biopsy
Description: A positive malignant residual mass was defined as focal 18F- Fluorothymidine (FLT) uptake within the residual mass greater than the normal mediastinal background uptake. FLT uptake within the mass lower than the mediastinal was considered non-malignant. The positive/negative FLT uptake was correlated with biopsy results within the residual mass (presence or absence of malignant tumor cells).
Time Frame: Up to 3.5 years
Population: 21/22 participants were analyzed because one participant was not treated ineligible per CT criteria. Data was collected for only the Arm/Group of participants with residual masses.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Scanned in the Evaluation of Residual Masses After Therapy: Patients undergo a 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F-18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scan to evaluate of a residual tumor mass after patients have completed therapy. Patients also undergo a biopsy or fine-needle aspiration, if clinically indicated.
  Biopsy: Biopsy taken [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans fine-needle aspiration: sample collected
Arm/Group | Participants Scanned in the Evaluation of Residual Masses After Therapy
Number analyzed (Participants) | 21
Participants
  Presence of FLT uptake | 9
  Absence of FLT uptake and FLT uptake lower than normal mediastinum | 12
  Positive Biopsy: number analyzed (Participants) | 11
  Positive Biopsy | 7
  Negative Biopsy: number analyzed (Participants) | 11
  Negative Biopsy | 4
  Biopsy not performed | 10
Statistical Analysis 1: Comparison: Participants Scanned in the Evaluation of Residual Masses After Therapy; Test type: Superiority; p < 0.001, Wilcoxon signed-rank test

2. Secondary Outcome: 18F- Fluorothymidine (FLT) Uptake Within the Tumor(s) Between Baseline vs Completion of Therapy Scans
Description: FLT uptake within the tumor(s) using standard uptake value (SUVmax) was compared between baseline and completion of therapy scans.
Time Frame: up to 4.5 years
Population: 8/9 participants were analyzed at baseline because the FLT dose failed synthesis in 1 participant. 6/9 participants were analyzed at completion of therapy because 1 participant refused to be imaged, 1 participant missed scan appointment, and 1 patient's FLT dose failed synthesis at baseline and was not scanned at completion of therapy either The rows at baseline and completion of therapy represent the pts: 8 patients were scanned at baseline and 6 pts were scanned at completion of therapy.
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- Participants Scanned at Baseline & After Chemotherapy: Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scans at baseline, after 2 courses of chemotherapy, and after completion of chemotherapy. Patients with residual FDG-positive mass after completion of therapy may be enrolled in group B.
  Fluordeoxyglucose F 18: Undergo scans
  [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans
  computed tomography: Undergo scans
Arm/Group | Participants Scanned at Baseline & After Chemotherapy
Number analyzed (Participants) | 8
SUVmax
  Baseline | 9.15 (2.84)
  Completion of therapy scans: number analyzed (Participants) | 6
  Completion of therapy scans | 0.9 (0.20)
Statistical Analysis 1: Comparison: Participants Scanned at Baseline & After Chemotherapy; Test type: Superiority; p = 0.0313, Wilcoxon matched-pairs signed rank test

3. Secondary Outcome: Tumor(s) Maximum Standard Uptake Value (SUVmax) at Baseline Scan and SUVmax After Completion Scan in Responders and Non-responders' Patients
Description: The SUVmax (defined as radiotracer uptake in a region of interest normalized by the injected activity and body weight) was measured within the tumor(s). The SUVmax was defined as the uptake value of the hottest pixels, within a volume of interest containing the entire tumor(s). SUVmax was calculated at baseline and after completion of therapy.
Time Frame: up to 4.5 years
Population: 8/9 participants were analyzed at baseline and 6/9 were analyzed after completion of therapy because 6 patients completed the 3 scans (baseline, at 2-cycles and after completion of therapy). This outcome measure data is collected only for one of the Arm/Group. The other group of participants were not scanned at baseline and after treatment. This data is for baseline (8 patients) and after therapy (6 patients). The outcome measure refers to baseline and after completion of therapy.
Measure: Median (Standard Deviation); unit: Standard Uptake Value (SUV) - units
Groups:
- Participants Scanned at Baseline & After Chemotherapy: Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scans at baseline, after 2 courses of chemotherapy, and after completion of chemotherapy. Fluorodeoxyglucose F 18: Undergo scans [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans
Arm/Group | Participants Scanned at Baseline & After Chemotherapy
Number analyzed (Participants) | 8
Standard Uptake Value (SUV) - units
  Baseline | 9.1 (2.8)
  After completion of scan: number analyzed (Participants) | 6
  After completion of scan | 1.5 (0.6)

4. Secondary Outcome: Tumor Uptake With Fluorothymidine (FLT) - Maximum Standard Uptake Value (SUVmax)
Description: The maximum standard uptake value (SUVmax) (defined as radiotracer uptake in a region of interest normalized by the injected activity and body weight) was measured within the tumor(s). The SUVmax was defined as the uptake value of the hottest pixels, within a volume of interest containing the entire tumor(s).
Time Frame: Up to 4.5 years
Population: 6/9 participants were analyzed after completion of therapy because the FLT dose failed synthesis in 1 participant at baseline and was not scanned at completion, 1 participant refused to be imaged and 1 participant missed scan appointment. The other group of participants were not scanned at baseline and after treatment.
Measure: Mean (Standard Deviation); unit: SUV
Groups:
- Participants Scanned at Baseline: Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scans at baseline. Fluorodeoxyglucose F 18: Undergo scans [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans
- Participants Scanned After Completion of Therapy: Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scans after completion of chemotherapy. Fluorodeoxyglucose F 18: Undergo scans [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans
Arm/Group | Participants Scanned at Baseline | Participants Scanned After Completion of Therapy
Number analyzed (Participants) | 6 | 6
SUV
  Patient 1: number analyzed (Participants) | 1 | 1
  Patient 1 | 10.9 | 0.9
  Patient 2: number analyzed (Participants) | 1 | 1
  Patient 2 | 4.8 | 1.0
  Patient 3: number analyzed (Participants) | 1 | 1
  Patient 3 | 10.3 | 1.3
  Patient 4: number analyzed (Participants) | 1 | 1
  Patient 4 | 9.1 | 0.9
  Patient 5: number analyzed (Participants) | 1 | 1
  Patient 5 | 9.3 | 0.6
  Patient 6: number analyzed (Participants) | 1 | 1
  Patient 6 | 9.2 | 0.9
  Group-level (at baseline and after completion of therapy) | 9.2 (1.9) | 0.9 (0.2)

5. Secondary Outcome: 18F-fluorodeoxyglucose (18FDG) Standardized Uptake Values (SUV) Estimated Maximum and Tumor: Blood Pool Ratio at 1-hour Post-injection
Description: After 1 hour post-injection of fluorodeoxyglucose (FDG), the maximum uptake value (SUVmax) (defined as radiotracer uptake in a region of interest normalized by the injected activity and body weight) was calculated was calculated within the residual mass. The ratio between SUVmax within the residual mass and SUVmean in the pool blood was measured.
Time Frame: up to 3.5 years
Population: 21/22 participants were analyzed because one participant was not treated ineligible per CT criteria. Data collected only from residual mass Group of patients for this Outcome Measure.
Measure: Number; unit: SUVmax/Tumor blood ratio
Arm/Group | Participants Scanned in the Evaluation of Residual Masses After Therapy
Number analyzed (Participants) | 21
SUVmax/Tumor blood ratio
  Patient 1: number analyzed (Participants) | 1
  Patient 1 | 4.6
  Patient 2: number analyzed (Participants) | 1
  Patient 2 | 8.4
  Patient 3: number analyzed (Participants) | 1
  Patient 3 | 10.1
  Patient 4: number analyzed (Participants) | 1
  Patient 4 | 3.8
  Patient 5: number analyzed (Participants) | 1
  Patient 5 | 6.9
  Patient 6: number analyzed (Participants) | 1
  Patient 6 | 6.7
  Patient 7: number analyzed (Participants) | 1
  Patient 7 | 5.4
  Patient 8: number analyzed (Participants) | 1
  Patient 8 | 4.7
  Patient 9: number analyzed (Participants) | 1
  Patient 9 | 4.6
  Patient 10: number analyzed (Participants) | 1
  Patient 10 | 10.3
  Patient 11: number analyzed (Participants) | 1
  Patient 11 | 4.8
  Patient 12: number analyzed (Participants) | 1
  Patient 12 | 3.8
  Patient 13: number analyzed (Participants) | 1
  Patient 13 | 4.0
  Patient 14: number analyzed (Participants) | 1
  Patient 14 | 6.9
  Patient 15: number analyzed (Participants) | 1
  Patient 15 | 6.4
  Patient 16: number analyzed (Participants) | 1
  Patient 16 | 15.8
  Patient 17: number analyzed (Participants) | 1
  Patient 17 | 11.2
  Patient 18: number analyzed (Participants) | 1
  Patient 18 | 2.1
  Patient 19: number analyzed (Participants) | 1
  Patient 19 | 3.8
  Patient 20: number analyzed (Participants) | 1
  Patient 20 | 3.5
  Patient 21: number analyzed (Participants) | 1
  Patient 21 | 9.1

6. Secondary Outcome: 3'-Deoxy-3'-[18F]-Fluorothymidine (FLT) Dynamic Influx Parameter (Ki) Standardized Uptake Values (SUV) Estimated Maximum at 1- and 2-hours Post-injection
Description: The maximum uptake value (SUVmax) (defined as radiotracer uptake in a region of interest normalized by the injected activity and body weight) was calculated within the residual mass at 1 h and at 2 hours post-injection of FLT.
Time Frame: up to 3.5 years
Population: This outcome measure was collected for Arm/Group of patients with residual tumor masses after therapy. 21/22 participants were analyzed in thisArm/Group because one participant was not scanned with FLT, ineligible per CT criteria. 18/21 were analyzed in the second Arm/Group because no scans were available for three participants at 2 hours post injection.
Measure: Mean (Standard Deviation); unit: SUV
Groups:
- Participants Scanned in the Evaluation of Residual Masses After Therapy at 1 Hour Post Injection: Participants with residual masses after therapy were evaluated with FLT-positron-emission tomography (PET)/computed tomography (CT), acquiring the images after 1 hour after the intravenous injection of FLT to evaluate the tumor uptake value at 1 hour post injection.
- Participants Scanned in the Evaluation of Residual Masses After Therapy at 2 Hours Post Injection: Participants with residual masses after therapy were evaluated with FLT-positron-emission tomography (PET)/computed tomography (CT), acquiring the images after 2 hours of the intravenous injection of FLT to evaluate the tumor uptake at at 2 hours post injection.
Arm/Group | Participants Scanned in the Evaluation of Residual Masses After Therapy at 1 Hour Post Injection | Participants Scanned in the Evaluation of Residual Masses After Therapy at 2 Hours Post Injection
Number analyzed (Participants) | 21 | 18
SUV
  Patient 1: number analyzed (Participants) | 1 | 1
  Patient 1 | 0.7 | NA — The 2 hour scan was not acquired.
  Patient 2: number analyzed (Participants) | 1 | 1
  Patient 2 | 2.0 | 1.8
  Patient 3: number analyzed (Participants) | 1 | 1
  Patient 3 | 8.9 | NA — The 2 hour scan was not acquired.
  Patient 4: number analyzed (Participants) | 1 | 1
  Patient 4 | 1.6 | 0.8
  Patient 5: number analyzed (Participants) | 1 | 1
  Patient 5 | 1.3 | 7.9
  Patient 6: number analyzed (Participants) | 1 | 1
  Patient 6 | 7.5 | 4.6
  Patient 7: number analyzed (Participants) | 1 | 1
  Patient 7 | 3.4 | 3.2
  Patient 8: number analyzed (Participants) | 1 | 1
  Patient 8 | 1.6 | 1.2
  Patient 9: number analyzed (Participants) | 1 | 1
  Patient 9 | 6.5 | 6.0
  Patient 10: number analyzed (Participants) | 1 | 1
  Patient 10 | 2.3 | 2.0
  Patient 11: number analyzed (Participants) | 1 | 1
  Patient 11 | 2.5 | 2.4
  Patient 12: number analyzed (Participants) | 1 | 1
  Patient 12 | 2.2 | 1.5
  Patient 13: number analyzed (Participants) | 1 | 1
  Patient 13 | 7.6 | 7.4
  Patient 14: number analyzed (Participants) | 1 | 1
  Patient 14 | 4.5 | 4.2
  Patient 15: number analyzed (Participants) | 1 | 1
  Patient 15 | 1.9 | 1.6
  Patient 16: number analyzed (Participants) | 1 | 1
  Patient 16 | 3.9 | 3.6
  Patient 17: number analyzed (Participants) | 1 | 1
  Patient 17 | 4.7 | 4.5
  Patient 18: number analyzed (Participants) | 1 | 1
  Patient 18 | 7.9 | 7.9
  Patient 19: number analyzed (Participants) | 1 | 1
  Patient 19 | 1.1 | 1.1
  Patient 20: number analyzed (Participants) | 1 | 1
  Patient 20 | 1.5 | NA — The 2 hour scan was not acquired.
  Patient 21: number analyzed (Participants) | 1 | 1
  Patient 21 | 6.4 | 5.4
  Overall participants | 3.6 (2.5) | 2.9 (2.0)

7. Secondary Outcome: Tumor(s) Maximum Standard Uptake Value (SUVmax) at Baseline and at Mid-treatment (Post-2 Cycles) Scan
Description: The SUVmax (defined as radiotracer uptake in a region of interest normalized by the injected activity and body weight) was measured within the tumor(s). The SUVmax was defined as the uptake value of the hottest pixels, within a volume of interest containing the entire tumor(s). SUVmax was calculated at baseline and after 2-cycles of therapy.
Time Frame: Up to 4.5 years
Population: 8/9 participants were analyzed because the FLT dose failed synthesis in 1 participant, 1 participant refused to be imaged.
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- Participants Scanned at Baseline, at 2 Cycles & After ChemotherapyChemotherapy: Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scans at baseline, after 2 courses of chemotherapy, and after completion of chemotherapy. Fluorodeoxyglucose F 18: Undergo scans [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans
Arm/Group | Participants Scanned at Baseline, at 2 Cycles & After ChemotherapyChemotherapy
Number analyzed (Participants) | 8
SUVmax
  Baseline | 9.15 (2.84)
  2-cycles post treatment | 1.5 (0.63)

8. Secondary Outcome: Time to Progression
Description: The time to progression (defined as time in months from 3'-deoxy-3'-[18F] fluorothymidine (FLT)-scan until patient progressed) was compared between the two groups (patients with higher Maximum Standard Uptake Value (SUVmax) vs lower SUVmax, using the median SUV value).
Time Frame: up to 4.5 years
Population: 3/6 participants were analyzed because 3 did not progress while on study. Data collected only from the Group of patients scanned at baseline and after chemotherapy for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Participants Scanned After Chemotherapy: Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scans after completion of chemotherapy. Patients with residual FDG-positive mass after completion of therapy may be enrolled in group B.
  Fluorodeoxyglucose F 18: Undergo scans [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans
Arm/Group | Participants Scanned After Chemotherapy
Number analyzed (Participants) | 3
Months | 18.29 (8.0)

9. Secondary Outcome: 18F- Fluorothymidine (FLT) Uptake, Positron-emission Tomography (PET) Standard Uptake Value (SUV)Max in Malignant Residual Tumors Versus Benign Lesions After Therapy
Description: FLT uptake was calculated within malignant residual tumors versus benign lesions using maximum standard uptake value (SUVmax).
Time Frame: up to 4.5 years
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- Participants Scanned in the Evaluation of Residual Masses After Therapy: Patients undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scans in the evaluation of FDG-positive residual masses after therapy. Patients also undergo a biopsy or fine-needle aspiration, if clinically indicated.
  Biopsy: Biopsy taken [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans fine-needle aspiration: sample collected
Arm/Group | Participants Scanned in the Evaluation of Residual Masses After Therapy
Number analyzed (Participants) | 21
SUVmax
  Malignant Lesions | 5.5 (2.2)
  Benign Lesions | 1.7 (0.6)

10. Other Pre Specified Outcome: Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 4 years, 7 months and 9 days.
Population: 8/9 patients were injected with the tracer (FLT) and scanned in the first Arm/Group, and 21/22 in the second Arm/Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Scanned at Baseline & After Chemotherapy | Participants Scanned in the Evaluation of Residual Masses After Therapy
Number analyzed (Participants) | 8 | 21
Participants | 7 | 20

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 4 years, 7 months and 9 days.
Description: 8/9 patients were injected with the tracer (FLT) and scanned in the first Arm/Group, and 21/22 in the second Arm/Group. The risk can only be for 8 patients and 21 participants who received FLT scan.
Groups:
- Participants Scanned in the Evaluation of Residual Masses After Therapy: Patients undergo a 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fluorodeoxyglucose F 18 (FDG) Positron-emission tomography (PET)/Computed tomography (CT) scan in the evaluation of FDG-positive residual masses after therapy. Patients also undergo a biopsy or fine-needle aspiration, if clinically indicated.
  Biopsy: Biopsy taken [3'-deoxy-3'-[F-18] fluorothymidine: Undergo scans computed tomography: Undergo scans fine-needle aspiration: sample collected
  fine-needle aspiration: sample collected
Arm/Group | Participants Scanned at Baseline & After Chemotherapy | Participants Scanned in the Evaluation of Residual Masses After Therapy
All-Cause Mortality (participants affected / at risk) | 3/8 | 5/21
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/21
Other Adverse Events (participants affected / at risk) | 1/8 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Scanned at Baseline & After Chemotherapy (N=8) | Participants Scanned in the Evaluation of Residual Masses After Therapy (N=21)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2013-03-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT00775268/Prot_SAP_000.pdf
  • Informed Consent Form: Early Response Consent (2013-02-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT00775268/ICF_001.pdf
  • Informed Consent Form: Residual Mass Consent (2013-02-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT00775268/ICF_002.pdf